CLINICAL TRIAL: NCT00446446
Title: Phase 2, Single-Arm, Open-Label, Multi-Center Trial of Second-Line Panitumumab Monotherapy in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: PRISM (Panitumumab Regimen In Second-line Monotherapy of Head and Neck Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20062088
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Cancer; Carcinoma; Head and Neck Cancer; Metastases; Metastatic Cancer; Metastatic or Recurrent Squamous Cell Carcinoma of Head and Neck; Oncology; Squamous Cell Carcinoma; Tumors
MeSH Terms: conditions — Neoplasms; Carcinoma; Head and Neck Neoplasms; Neoplasm Metastasis; Carcinoma, Squamous Cell | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental): articipants received panitumumab as an intravenous infusion at a dose of 9 mg/kg every 21 days until disease progression, unacceptable toxicity, withdrawal of consent, death, or end of study.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Panitumumab was administered over a 1 hour intraveneous (IV) infusion at a dose of 9 mg/kg every 21 days.
  Other Names: Vectibix

SUMMARY:
To estimate the effect of second-line panitumumab monotherapy on objective response in patients with metastatic or recurrent squamous cell carcinoma of head and neck (SCCHN).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of head and neck (SCCHN) of oropharynx, oral cavity, hypopharynx, or larynx with at least 1 measurable lesion using computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Diagnosis of recurrent disease determined to be incurable by surgery or radiotherapy
* Karnofsky Performance Status (KPS) score ≥ 60% at screening
* Men or women age ≥18 years
* Adequate hematologic, electrolyte and hepatic functions and negative pregnancy test

Exclusion Criteria:

* Subject received > 1 chemotherapy regimen for the treatment of metastatic or recurrent disease
* Concomitant chemotherapy for recurrent disease administered solely for the purpose of radiation sensitization during re-irradiation will not be counted towards this chemotherapy regimen
* Nasopharyngeal carcinoma, salivary gland and primary skin SCCHN, or symptomatic central nervous system (CNS) metastases
* History of interstitial lung disease, significant cardiovascular disease, or another primary cancer
* Known positive test for human immunodeficiency virus (HIV) infection, hepatitis C virus, acute or chronic hepatitis B infection
* Known allergy or hypersensitivity to any component of panitumumab
* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy (eg, panitumumab, cetuximab) or treatment with small molecule EGFr inhibitors (eg, gefitinib, erlotinib, lapatinib) for recurrent or metastatic disease with the following exceptions:

  * Prior EGFr inhibitor therapy is allowed if received as part of prior multimodality treatment (eg, as radiation sensitizer) and completed > 24 weeks prior to randomization
  * Subjects who received no more than one dose of cetuximab and discontinued prior to progression due to documented severe infusion reaction are eligible.
* Significant thromboembolic event ≤ 8 weeks prior to enrollment
* Subjects not recovered from all previous acute radiotherapy-related toxicities
* History of severe skin disorder that in the opinion of the investigator may interfere with study conduct
* History of any medical, or psychiatric condition, or laboratory abnormality that may interfere with the interpretation of study results
* Subject is currently in a clinical trial ≤ 30 days prior to enrollment
* Subjects requiring use of immunosuppressive agents however corticosteroids are allowed
* Man or woman of child-bearing potential who do not consent to use adequate contraceptive precautions during the course of the study
* Female subject who is pregnant or breast-feeding
* Subject requiring major surgery using general/spinal anesthesia ≤ 28 days prior to enrollment, or minor surgery ≤ 14 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10-30 (Actual); Primary Completion 2010-12-15 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Rischin D, Spigel DR, Adkins D, Wein R, Arnold S, Singhal N, Lee O, Murugappan S. PRISM: Phase 2 trial with panitumumab monotherapy as second-line treatment in patients with recurrent or metastatic squamous cell carcinoma of the head and neck. Head Neck. 2016 Apr;38 Suppl 1:E1756-61. doi: 10.1002/hed.24311. Epub 2015 Dec 17. PMID 26681429
- [Background] Spigel D. Second-line panitumumab monotherapy for treatment of advanced head and neck cancer: the PRISM Trial. Community Oncology. 2008;5(Supp 11):1-4.
- [Background] Kim TW, Elme A, Park JO, Udrea AA, Kim SY, Ahn JB, Valencia RV, Krishnan S, Manojlovic N, Guan X, Lofton-Day C, Jung AS, Vrdoljak E. Final Analysis of Outcomes and RAS/BRAF Status in a Randomized Phase 3 Study of Panitumumab and Best Supportive Care in Chemorefractory Wild Type KRAS Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2018 Sep;17(3):206-214. doi: 10.1016/j.clcc.2018.03.008. Epub 2018 Mar 21. PMID 29703606
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 patients with metastatic or recurrent squamous cell carcinoma of the head and neck were screened of whom 52 were enrolled at 22 study centers in North America (20 study centers) and Australia (2 study centers) between October 2007 and December 2009.
Pre-assignment Details: Results are reported for the primary analysis with a data cut-off date of 16 December 2010.
Groups:
- Panitumumab: Participants received panitumumab as an intravenous infusion at a dose of 9 mg/kg every 21 days until disease progression, unacceptable toxicity, withdrawal of consent, death, or end of study.
Period: Overall Study
Arm/Group | Panitumumab
Started | 52
Completed | 28 (Participants who completed the 60-day safety visit)
Not Completed | 24
Not completed — Death | 10
Not completed — Withdrawal by Subject | 6
Not completed — Other | 4
Not completed — Disease Progession | 2
Not completed — Adverse Event | 1
Not completed — On Treatment at Time of Data Cut-off | 1

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 48
  Black or African American | 3
  Other | 1
Primary Tumor Site [Number; unit: participants]
  Oropharynx | 18
  Hypopharynx | 1
  Larynx | 13
  Oral Cavity | 20
Cancer Stage of Diagnosis [Number; unit: participants]
  Locally recurrent disease without metastases | 11
  Metastatic | 41
Prior Treatment for Head and neck Cancer [Number; unit: participants] — Participants may have received more than one prior treatment.
  participants
    Prior chemotherapy | 52
    Prior radiotherapy | 48
    Prior surgery | 46
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction;
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  2. = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours;
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  4. = Completely disabled, confined to bed or chair;
  5. = Dead.
  participants
    0 = (Fully Active) | 20
    1 = (Restrictive but Ambulatory) | 31
    2 = (Ambulatory unable to Work) | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Assessments are based on investigator's review of scans using a modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Objective response rate was defined as the percentage of participants with a best tumor response of complete response (CR) or partial response (PR) prior to initiation of subsequent anti-cancer therapy. CR or PR was confirmed no less than 28 days after the criteria for response were first met. CR: Disappearance of all target lesions, non-target lesions and no new lesions. PR: At least a 30% decrease in the size of target lesions and no progression of existing non-target lesions (defined as an increase in lesion size of ≥ 20%) and no new lesions, or, the disappearance of all target lesions and the persistence of one or more non-target lesion(s) not qualifying for either CR or progressive disease (PD) and no new lesions.
Time Frame: From first dose of study drug until the data cut-off date of 16 December 2010. Median duration of treatment was 9.0 weeks (range: 3.0 to 68.9 weeks).
Population: Full analysis set (all enrolled participants who received at least 1 dose of panitumumab) with measurable disease at Baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
percentage of participants | 3.9 [0.5 to 13.5]

2. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from Study Day 1 to the first CR or PR that was subsequently confirmed.
Time Frame: From first dose until the data cut-off date of 16 December 2010; median duration of treatment was 9.0 weeks (range: 3.0 to 68.9 weeks)
Population: Full analysis set participants with objective responses
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 2
weeks | 14.3 [4.9 to 23.7]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from first confirmed CR or PR to the earliest date of disease progression per a modified version of the RECIST criteria (version 1.0). Participants not meeting the criteria for progression by the analysis data cut-off date were censored at the date of last evaluable disease assessment. Duration of response was analyzed using the Kaplan-Meier method.
  PD: At least a 20% increase in the size of target lesions, or an increase of 20% or greater of non-target lesions and the lesion(s) measure ≥ 10 mm in one dimension at the time of progression, or any new lesions.
Time Frame: as for outcome 2
Population: Full analysis set participants with an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 2
months | NA [NA to NA] — Duration of response could not be estimated due to the low number of events at the time of data cut-off.

4. Secondary Outcome: Rate of Disease Control
Description: Rate of disease control was defined as the percentage of participants with CR, PR, or stable disease (SD), as defined by a modified version of the RECIST criteria (version 1.0), prior to initiation of subsequent anti-cancer therapy.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD of target lesions and no progression of non-target lesions and no new lesions, or, if no target lesions were identified at screening, the persistence of one or more non-target lesion(s) not qualifying for either CR or PD.
Time Frame: as for outcome 2
Population: Full analysis set with measurable disease at Baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
percentage of participants | 39.2 [25.8 to 53.9]

5. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from Day 1 to the date of disease progression using a modified version of the RECIST criteria (version 1.0). Participants not meeting the criteria for progression by the analysis data cut-off date were censored at the date of last evaluable disease assessment. Time to progression was analyzed using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 52
months | 1.4 [1.3 to 2.4]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from Day 1 to the first date of disease progression, as defined by a modified version of the RECIST criteria (version 1.0), or death due to any cause (whichever comes first). Participants who were alive who did not meet the criteria for progression by the analysis data cut-off date were censored at the date of last evaluable disease assessment.
  PFS was analyzed using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 52
months | 1.4 [1.3 to 2.4]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from Day 1 to the date of death. For participants who did not die while on study, or were lost to follow-up, survival was censored at the end of study, or the date of last contact (whichever was first).
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 52
months | 5.1 [4.3 to 8.3]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event (AE) was graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (where grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening and grade 5=fatal) with the exception of some dermatology/skin AEs that were graded using the CTCAE v3.0 with modifications. Serious AEs include any event that was fatal, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or other significant medical hazard. Treatment-related adverse events (TRAEs) are those for which the investigator considered there to be a reasonable possibility that the event may have been caused by study drug.
Time Frame: The reporting time frame for Adverse Events is from first dose date to 30 days since the last dose date date. The median time frame is 2.4 months.
Population: Safety analysis set (all enrolled participants who received at least 1 dose of panitumumab)
Measure: Number; unit: participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 52
participants
  Any adverse event | 52
  Worst grade of 3 | 18
  Worst grade of 4 | 4
  Worst grade of 5 | 5
  Serious adverse event | 14
  Leading to discontinuation of panitumumab | 4
  Leading to removal from study | 5
  Treatment-related adverse event | 45
  Treatment-related worst grade of 3 | 9
  Treatment-related worst grade of 4 | 1
  Treatment-related worst grade of 5 | 1
  Serious treatment-related adverse event | 3
  TRAE leading to discontinuation of panitumumab | 0
  Treatment-related leading to removal from study | 2

ADVERSE EVENTS:
Time Frame: The reporting time frame for Adverse Events is from first dose date to 30 days since the last dose date date. The median time frame is 2.4 months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Panitumumab
Serious Adverse Events (participants affected / at risk) | 14/52
Other Adverse Events (participants affected / at risk) | 50/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=52)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
VISION BLURRED (Eye disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 2
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 2
ASTHENIA (General disorders) | 1
FATIGUE (General disorders) | 1
PAIN (General disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
BRONCHITIS (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=52)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3
CONSTIPATION (Gastrointestinal disorders) | 7
DIARRHOEA (Gastrointestinal disorders) | 8
DYSPHAGIA (Gastrointestinal disorders) | 4
NAUSEA (Gastrointestinal disorders) | 7
ORAL PAIN (Gastrointestinal disorders) | 3
VOMITING (Gastrointestinal disorders) | 5
FATIGUE (General disorders) | 16
MUCOSAL INFLAMMATION (General disorders) | 4
PAIN (General disorders) | 4
PARONYCHIA (Infections and infestations) | 3
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 3
WEIGHT DECREASED (Investigations) | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 7
DEHYDRATION (Metabolism and nutrition disorders) | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
INSOMNIA (Psychiatric disorders) | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 12
DRY SKIN (Skin and subcutaneous tissue disorders) | 11
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 8
RASH (Skin and subcutaneous tissue disorders) | 27
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 4
SWELLING FACE (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.